CLINICAL TRIAL: NCT03278834
Title: The Use of Neuromuscular Electrical Stimulation With Pelvic Fracture Rehabilitation: A Randomised, Double Blind, Pilot Study
Brief Title: NMES and Pelvic Fracture Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NMES Pilot Study
Record Dates: First submitted 2017-07-13; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-07

CONDITIONS: Trauma; Rehabilitation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Treatment and intervention group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Neuromuscular muscle stimulation machine - Muscle stimulation machine to be used on glutes and abductors on disuse atrophy setting.
  Twice per day for 45 minutes.
  Exercise - Home exercises programme once per day with 10 exercises.
  Interventions: Device: Neuromuscular muscle stimulation machine- Strength Setting
- Placebo Group (Placebo Comparator): Neuromuscular muscle stimulation- Muscle stimulation machine to be used on glutes and abductors on TENS setting. Twice per day for 45 minutes.
  Exercise - Home exercises programme once per day with 10 exercises.
  Interventions: Device: Neuromuscular muscle stimulation machine - TENS Setting

INTERVENTIONS:
Device: Neuromuscular muscle stimulation machine- Strength Setting — Muscle stimulation to strength skeletal muscle
  Arms: Intervention Group
Device: Neuromuscular muscle stimulation machine - TENS Setting — Muscle stimulation to mimic the intervention but without the strength gains.
  Arms: Placebo Group

SUMMARY:
Objectives: The acute care of pelvic fractures has improved recently however there are no formal guidelines for rehabilitation of these types of fractures. Patients have long periods of non-weight bearing causing muscle wastage. Neuromuscular electrical stimulation (NMES) has proven to minimise muscle loss. However, this has not previously been investigated within this patient population.

Design: Double blind, randomised, feasibility study.

Setting: NHS trust hospital setting.

Participants: Nine patients with surgically fixed pelvic fractures were randomly allocated at six weeks post fracture.

Interventions: The intervention group completed six weeks of NMES. The placebo group used transcutaneous electrical nerve stimulation (TENS).

Main outcome measures: Peak torque (Nm) was calculated in the operated limb at 12 weeks using the non-operated limb as a baseline. Compliance and intensity levels were recorded. Feasibility of NMES was evaluated using a feasibility questionnaire. Pain was measured at six and 12 weeks using a visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were any patient with a pelvic fracture that was surgically fixed with no associated injuries and able to give written informed consent.
* Pelvic fractures including acetabular and pelvic ring fracture that were fixed using open reduction internal fixation (ORIF) were considered.

Exclusion Criteria:

* Exclusion criteria were patients who could not comply with the NMES or who had previous mental health diagnosis.
* Patients who may be pregnant, have severe kidney injury or have a pacemaker were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 12 weeks post operation
  Peak Torque muscle strength

SECONDARY OUTCOMES:
Feasibility questionnaire | 12 weeks post operation
  questionnaire of 10 questions